CLINICAL TRIAL: NCT00089050
Title: A Phase II Trial Combining Gemtuzumab Ozogamicin (Mylotarg) With Cyclosporine for the Treatment of Relapsed Acute Myeloid Leukemia in Adults Over Age 60
Brief Title: Gemtuzumab Ozogamicin and Cyclosporine in Treating Older Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1820.00; FHCRC-1820.00; CDR0000378021 (Registry Identifier: PDQ)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Congenital Abnormalities | interventions — Cyclosporine; Gemtuzumab

INTERVENTIONS:
Drug: cyclosporine
Drug: gemtuzumab ozogamicin

SUMMARY:
RATIONALE: Monoclonal antibodies such as gemtuzumab ozogamicin can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Cyclosporine may increase the effectiveness of gemtuzumab ozogamicin by making cancer cells more sensitive to the drug. Combining gemtuzumab ozogamicin with cyclosporine may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving gemtuzumab ozogamicin together with cyclosporine works in treating older patients with relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of gemtuzumab ozogamicin and cyclosporine, in terms of the complete remission rate, in older patients with relapsed acute myeloid leukemia.
* Determine the toxicity and pharmacokinetics of this regimen in these patients.

Secondary

* Correlate clinical response with laboratory studies of drug susceptibility in patients treated with this regimen.

OUTLINE: Patients receive cyclosporine IV continuously over 72 hours on days 1-3 and 15-17. Eight hours after initiation of each cyclosporine infusion, patients receive gemtuzumab ozogamicin IV over 2 hours on days 1 and 15. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 25-50 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed acute myeloid leukemia (AML) by bone marrow aspirate

  * More than 20% blasts by morphologic criteria
  * Relapsed disease ≥ 3 months after prior complete remission
* Blasts CD33-positive by flow cytometry
* No primary hematologic disorder that preceded initial presentation with AML
* No documented secondary AML related to prior chemotherapy or toxin exposure
* No acute promyelocytic leukemia (FAB M3)
* Not a candidate for transplant therapy
* No active CNS leukemia

PATIENT CHARACTERISTICS:

Age

* 60 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC ≤ 30,000/mm^3 (hydroxyurea allowed)

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* HIV negative
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not planning hematopoietic stem cell transplantation immediately after study therapy

Chemotherapy

* See Disease Characteristics
* See Hematopoietic

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 1 month since prior investigational agents
* No other concurrent anticancer therapy
* No administration of any of the following for 24 hours after cyclosporine administration:

  * Diltiazem
  * Verapamil
  * Erythromycin
  * Clarithromycin
  * Metoclopramide
  * Phenytoin
  * Rifampin
  * Phenobarbital
  * Aminoglycosides
  * Amphotericin B
  * Vancomycin
  * Cimetidine
  * Ranitidine
  * Trimethoprim/sulfamethoxazole
  * Ketoconazole
  * Fluconazole
  * Itraconazole
  * Voriconazole
  * Carbamazepine

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of complete remission rate
Toxicity
Pharmacokinetics

SECONDARY OUTCOMES:
Correlate clinical response to laboratory studies of drug susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H. Petersdorf, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States